CLINICAL TRIAL: NCT05886387
Title: Effect of Intraoperative PEEP With Recruitment Manoeuvres on the Occurrence of Postoperative Pulmonary Complications During General Anaesthesia--a Bayesian Analysis of Three Randomised Clinical Trials of Intraoperative Ventilation
Brief Title: a Bayesian Analysis of Three Randomised Clinical Trials of Intraoperative Ventilation
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Hospital Israelita Albert Einstein (Other); University Hospital Carl Gustav Carus (Other); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: Bayes_Repeat
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Mechanical Ventilation Complication; Surgery; Pulmonary Complication; Postoperative Complications
Keywords: Mechanical ventilation,; Bayesian analysis; PEEP; Recruitment Maneuvers; Intraoperative Mechanical Ventilation; Postoperative complications; Perioperative medicine
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High PEEP + Recruitment Maneuvers: Patients who received intraoperatively high PEEP (10-12 cmH2O) after a recruitment maneuvers as per the original study protocol
  Interventions: Other: High PEEP + Recruitment maneuvers
- Standard PEEP: Patients who received intraoperatively standard PEEP (0-5 cmH2O) without recruitment maneuvers
  Interventions: Other: Standard PEEP. Low positive end-expriatory pressure

INTERVENTIONS:
Other: High PEEP + Recruitment maneuvers — The use of a High PEEP (positive end-expiratory pressure) level after recruiting collapsed alveoli can protect from mechanical ventilation associated lung injury
  Groups: High PEEP + Recruitment Maneuvers
Other: Standard PEEP. Low positive end-expriatory pressure — Mechanical ventilation is managed with a low standard PEEP without recruitment manneuvers
  Groups: Standard PEEP

SUMMARY:
The investigators designed a protocol for a Bayesian unplanned posthoc analysis using the pooled dataset from three large randomized clinical trials. The primary endpoint will be a composite of postoperative pulmonary complications (PPC) within the first seven postoperative days, which reflects the primary endpoint of the original studies. The investigators will carry out a reanalysis of the harmonised database using Bayesian statistics.

DETAILED DESCRIPTION:
Background: Using the frequentist approach, a recent meta-analysis of three randomized clinical trials in patients undergoing intraoperative ventilation during general anesthesia for major surgery. failed to show the benefit of ventilation that uses high positive end expiratory pressure with recruitment maneuvers when compared to ventilation that uses low positive end-expiratory pressure without recruitment maneuvers.

Methods: The investigators designed a protocol for a Bayesian analysis using the pooled dataset. The multilevel Bayesian logistic model will use the individual patient data. Prior distributions will be prespecified to represent a varying level of skepticism for the effect estimate. The primary endpoint will be a composite of postoperative pulmonary complications (PPC) within the first seven postoperative days, which reflects the primary endpoint of the original studies. The investigators preset a range of practical equivalence to assess the futility of the intervention with an interval of odds ratio (OR) between 0.9 and 1.1 and assess how much of the 95% of highest density interval (HDI) falls between the region of practical equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Planned for major surgery
* At risk for pulmonary complications

Exclusion Criteria:

* Planned thoracic surgery .
* Unscheduled surgery (i.e., urgent, or emergent surgeries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing mechanical ventilation for general anesthesia for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 3836 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative pulmonary complications | Until day seven or hospital discharge, whichever comes first ]

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- IRCCS San Martino Policlinico Hospital, Genoa, Italy
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- See also: Association between ventilation parameter and postoperative complications — https://pubmed.ncbi.nlm.nih.gov/31157366/
- See also: PROBESE Study — https://pubmed.ncbi.nlm.nih.gov/26947624/
- See also: iPRVE study — https://pubmed.ncbi.nlm.nih.gov/29371130/
- See also: PROVHILO study — https://pubmed.ncbi.nlm.nih.gov/24894577/
- See also: The Association of Intraoperative driving pressure with postoperative pulmonary complications in open versus closed abdominal surgery patients — https://pubmed.ncbi.nlm.nih.gov/33740885/